CLINICAL TRIAL: NCT00458783
Title: Red Cell Storage Duration and Outcomes in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 07-140
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Blood Transfusion; Cardiac Surgery
Keywords: Transfusion; Cardiac; Blood storage duration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolonged RBC storage (Active Comparator): Transfusion with oldest available matching RBCs.
  Interventions: Biological: Prolonged RBC storage
- Short RBC storage (Active Comparator): Transfusion with youngest available matching RBCs.
  Interventions: Biological: Short RBC storage

INTERVENTIONS:
Biological: Prolonged RBC storage — Transfusion with oldest available matching RBCs
  Arms: Prolonged RBC storage
Biological: Short RBC storage — Transfusion with youngest available matching RBCs
  Arms: Short RBC storage

SUMMARY:
The purpose of this study is to determine whether length of storage of RBC is related to postoperative morbid outcomes in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Subjects undergoing cardiac surgery will be randomized into one of two groups. Group A will receive transfused blood that has storage duration less than 14 days. Group B will receive transfused blood with a storage duration of more than 20 days.

ELIGIBILITY:
Inclusion Criteria:

* All primary and reoperative adult cardiac surgical patients undergoing cardiopulmonary bypass for coronary artery bypass grafting, coronary artery bypass grafting with a valve procedure, isolated valve procedures, ascending aortic aneurysm or dissection repair alone or combined with CABG and valve procedures

Exclusion Criteria:

* Age less than 18 years
* Descending thoracic aortic aneurysm repairs
* Left or right ventricular assist devices
* Those unable to receive blood for religious reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3942 (Actual)
Dates: Start 2007-04; Primary Completion 2018-12 (Actual); Study Completion 2019-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andra Duncan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kekre N, Mallick R, Allan D, Tinmouth A, Tay J. The impact of prolonged storage of red blood cells on cancer survival. PLoS One. 2013 Jul 16;8(7):e68820. doi: 10.1371/journal.pone.0068820. Print 2013. PMID 23874777

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From July 2007 to May 2016, 3942 adults undergoing coronary artery bypass grafting, cardiac valve procedures, or ascending aorta repair, either alone or in combination were enrolled in the study. 3835 adults were randomized to transfusion of RBCs stored for ≤ 14 days (younger units) or for ≥ 20 days (older units) intraoperatively and throughout the postoperative hospitalization
Period: Overall Study
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Started | 1914 | 1921
Completed | 686 | 701
Not Completed | 1228 | 1220
Not completed — Protocol Violation | 1228 | 1220

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolonged RBC Storage | Short RBC Storage | Total
Number analyzed (Participants) | 686 | 701 | 1387
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (12) | 69 (12) | 69 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 326 | 381 | 707
  Male | 360 | 320 | 680
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 28 (5.9) | 28 (5.9) | 28 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Primary Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Morbid Outcomes in Patients Undergoing Cardiac Surgery.
Description: The primary composite endpoint was the occurrence of mortality or multisystem organ failure, cardiac events (ventricular tachycardia, fibrillation, or asystole; atrial fibrillation), pulmonary events (pneumonia, prolonged postoperative ventilation, pulmonary embolus), neurologic events (stroke, coma), renal failure, infection (deep sternal wound infection, sepsis), gastrointestinal events (ischemia, infarction), any reoperation (for bleeding, tamponade, cardiac dysfunction), and vascular events (dissection, limb ischemia), as defined for the STS database.
Time Frame: 30 days post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 360 | 362
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; p = 0.08, generalized estimating equation (GEE); Generalized estimating equation (GEE) distinct-effects model; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.50 to 1.2]

2. Primary Outcome: Effect of RBC Age on Occurrence of Mortality or Multisystem Organ Failure Events
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Mortality or Multisystem Organ Failure events in Patients Undergoing Cardiac Surgery.
Time Frame: 30 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 24 | 16
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; Odds Ratio, log = 0.64, 95% CI 2-sided [0.25 to 1.6]

3. Primary Outcome: Effect of RBC Age on Occurrence of Neurologic Events
Description: Neurologic events includes stroke and coma. Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Mortality or Neurologic events in Patients Undergoing Cardiac Surgery.
Time Frame: 30 days post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 19 | 14
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; Odds Ratio, log = 0.72, 95% CI 2-sided [0.26 to 2.0]

4. Primary Outcome: Effect of RBC Age on Occurrence of Pulmonary Events.
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Pulmonary events in Patients Undergoing Cardiac Surgery.
  Pulmonary events include pneumonia, prolonged postoperative ventilation and pulmonary embolus.
Time Frame: 30 days post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 113 | 106
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; Odds Ratio, log = 0.90, 95% CI 2-sided [0.59 to 1.4]

5. Primary Outcome: Effect of RBC Age on Occurrence of Renal Failure
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Renal Failure in Patients Undergoing Cardiac Surgery.
Time Frame: 30 days post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 36 | 32
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; Odds Ratio, log = 0.86, 95% CI 2-sided [0.43 to 1.8]

6. Primary Outcome: Effect of RBC Age on Occurrence of Infection Events
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Infection events in Patients Undergoing Cardiac Surgery.
  Infection events include deep sternal wound infection and sepsis.
Time Frame: 30 days post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 12 | 10
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; Risk Ratio, log = 0.81, 95% CI 2-sided [0.24 to 2.8]

7. Primary Outcome: Effect of RBC Age on Occurrence of Atrial Fibrillation
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Atrial fibrillation in Patients Undergoing Cardiac Surgery.
Time Frame: 30 days post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 238 | 258
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; Odds Ratio, log = 1.10, 95% CI 2-sided [0.80 to 1.5]

8. Primary Outcome: Effect of RBC Age on Occurrence of Asystole
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Asystole in Patients Undergoing Cardiac Surgery.
Time Frame: 30 days post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 29 | 13
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; Odds Ratio, log = 0.43, 95% CI 2-sided [0.16 to 1.1]

9. Primary Outcome: Effect of RBC Age on Occurrence of Gastrointestinal Events
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Gastrointestinal events in Patients Undergoing Cardiac Surgery.
  Gastrointestinal events include ischemia and infarction.
Time Frame: 30 days post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 33 | 28
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; Odds Ratio, log = 0.82, 95% CI 2-sided [0.39 to 1.7]

10. Primary Outcome: Effect of RBC Age on Occurrence of Any Reoperation
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to any Postoperative Reoperation in Patients Undergoing Cardiac Surgery.
  Reoperation for bleeding, tamponade and cardiac dysfunction.
Time Frame: 30 days post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 81 | 69
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; Odds Ratio, log = 0.82, 95% CI 2-sided [0.50 to 1.3]

11. Primary Outcome: Effect of RBC Age on Occurrence of Vascular Events
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Vascular events in Patients Undergoing Cardiac Surgery.
  Vascular events include dissection and limb ischemia.
Time Frame: 30 days post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Participants | 9 | 7
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; Odds Ratio, log = 0.76, 95% CI 2-sided [0.18 to 3.2]

12. Secondary Outcome: Effect of RBC Age on Intensive Care Unit (ICU) Length of Stay.
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Intensive Care Unit (ICU) Length of Stay in Patients Undergoing Cardiac Surgery.
Time Frame: The total hours from start to end in the Intensive Care Unit (ICU).
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Hours | 54 [29 to 114] | 51 [28 to 113]
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; p = 0.9, Regression, Cox; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.94 to 1.29] — The 95%CI is interim adjusted

13. Secondary Outcome: Effect of RBC Age on Postoperative Hospital Lengths of Stay.
Description: Aim is to Determine Whether Length of Storage of Red Blood Cells is Related to Postoperative Hospital Lengths of Stay in Patients Undergoing Cardiac Surgery.
Time Frame: The total days from start to end of the Hospital Stay.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Prolonged RBC Storage | Short RBC Storage
Number analyzed (Participants) | 686 | 701
Days | 9 [7 to 13] | 9 [7 to 13]
Statistical Analysis 1: Comparison: Prolonged RBC Storage vs Short RBC Storage; Test type: Superiority; p = 0.07, Regression, Cox; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.85 to 1.18] — The 95%CI is interim adjusted

ADVERSE EVENTS:
Time Frame: 30 days post surgery.
Arm/Group | Prolonged RBC Storage | Short RBC Storage
All-Cause Mortality (participants affected / at risk) | 23/686 | 15/701
Serious Adverse Events (participants affected / at risk) | 360/686 | 362/701
Other Adverse Events (participants affected / at risk) | 0/686 | 0/701
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prolonged RBC Storage (N=686) | Short RBC Storage (N=701)
Multisystem organ failure (General disorders) | 3 | 3
Stroke (Nervous system disorders) | 6 | 7
Coma (Nervous system disorders) | 14 | 9
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Prolonged ventilation (Respiratory, thoracic and mediastinal disorders) | 107 | 99
Renal morbidity (Renal and urinary disorders) | 36 | 32
Deep sternal wound infection (Infections and infestations) | 2 | 3
Septicemia/sepsis (Immune system disorders) | 10 | 7
Atrial fibrillation (Cardiac disorders) | 238 | 258
Asystole (Cardiac disorders) | 29 | 13
Gastrointestinal morbidity (Gastrointestinal disorders) | 33 | 28
Bleeding/tamponade (Surgical and medical procedures) | 44 | 36
Graft occlusion/valve dysfunction, noncardiac reasons (Surgical and medical procedures) | 47 | 41
Aortic or femoral artery dissection (Vascular disorders) | 1 | 0
Acute limb ischemia (Vascular disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-05-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT00458783/Prot_SAP_000.pdf